CLINICAL TRIAL: NCT06575647
Title: Mass Drug Administration of Tafenoquine for P. Vivax Radical Cure: Safety and Feasibility Study
Brief Title: Vivax Elimination With Tafenoquine (VET) Study
Acronym: VET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shoklo Malaria Research Unit (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAL24004
Record Dates: First submitted 2024-08-19; First posted 2024-08-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Malaria; Malaria, Vivax; Plasmodium Vivax; Plasmodium Vivax Malaria
Keywords: Mass drug administration; Plasmodium Vivax Malaria; Tafenoquine; Malaria elimination; Chloroquine prophylaxis
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — tafenoquine

STUDY DESIGN:
Intervention Model Description: Cross-sectional study with safety and feasibility assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tafenoquine (Experimental): Tafenoquine KODATEF® 100 mg film-coated tablets will be purchased from Biocelect (Suite 5.02, Level 5, 139 Macquarie Street, Sydney NSW, 2000 Australia).
  Tafenoquine will be given as follows,
  >10 kg to ≤ 20 kg - 150 mg (1 tab), >20 kg to ≤ 35 kg - 300 mg (2 tabs), > 35 kg - 450 mg (3 tabs)
  Interventions: Drug: Tafenoquine

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine KODATEF® 100 mg film-coated tablets will be purchased from Biocelect (Suite 5.02, Level 5, 139 Macquarie Street, Sydney NSW, 2000 Australia).
  Tafenoquine will be given as follows,
  >10 kg to ≤ 20 kg - 150 mg (1 tab), >20 kg to ≤ 35 kg - 300 mg (2 tabs), > 35 kg - 450 mg (3 tabs)

SUMMARY:
Theoretically, so long as there is a sink-source for malaria, transmission could be sustained at very low level (even at sub-microscopic oscillation) and reintroduce malaria either as sporadic cases or as resurgent outbreak. Uncertainty or shortage in financing has typically limited the malaria control or elimination projects to go further beyond the "Pre-elimination phase". Since malaria is no longer a top scoring mortality in national statistics in South East Asia, the governments/stakeholders are less willing to allocate from the austerity budget. There are proven evidence of resurgences after cessation of intervention programs where over 90% of all resurgence events were attributed to the interruption of malaria control programmes. In Karen state Myanmar-Thailand border, multiple factors including a cascade of political, financial, and logistical fiascos have compounded on the ongoing malaria elimination activities. Deleterious impacts after military coup since 2021 February including cessation of foreign investment, humanitarian aids, Civil Dis-obedience Movement of government staff and resuming armed-conflicts have strained the nearly failed health infrastructure of the country to a collapse stage. Interruption of the National Malaria Control activities due to the health system failure and accelerating combats countrywide could inevitably lead to the overturn in recently achieved malaria pre-elimination status especially in Karen state.

The disruption in health services within Myanmar is already resulting in an increase in malaria. Supply of the first line antimalarial drug artemether-lumefantrine, and other essential malaria control interventions, has been interrupted. The study is proposed to evaluate the impact of Mass Drug Administration (MDA) in 3 villages in Karen state with consistently high incidence of P. vivax and spatially clustered within 5 km radius. This proposal outlines a study to assess the feasibility and the safety of tafenoquine MDA.

DETAILED DESCRIPTION:
Malaria remains a major health concern in Myanmar, particularly in Karen State along the Myanmar-Thailand border, where disruptions in health services have led to a significant increase in cases. To address this, a study is proposed to assess the feasibility and safety of Mass Drug Administration (MDA) using tafenoquine, a single-dose treatment for P. vivax malaria, which has been approved in several countries, including Thailand. The study will focus on three high-incidence villages in Karen State, Myanmar, with a total population of around 1,000.

In this study, the entire village population will be screened for malaria using Rapid Diagnostic Tests (RDT) and PCR, a highly sensitive method that detects parasites by copying and identifying their unique genetic material in blood samples. Participants who test positive for malaria by RDT will receive standard treatment. Additionally, all participants will be screened for their G6PD enzyme status and will receive tafenoquine if G6PD levels are above 6.0 units, or chloroquine prophylaxis if their enzyme levels are lower or if they are pregnant. Impact of MDA on reduction in malaria incidence by RDT and prevalence by PCR will also be evaluated as a secondary outcome of the study.

Participation is voluntary, and participants can withdraw at any time. They will receive full information about the study's risks and benefits before deciding whether to participate.

Risks:

According to previous research conducted both in this context and in other regions, tafenoquine and chloroquine are generally safe, with side effects usually being mild. The most common side effects are nausea and mild to moderate abdominal pain. A research team led by a medical doctor will be on hand to manage any side effects, and a referral system will be established in case of any serious adverse events.

Benefits:

If successful, the study could significantly reduce malaria cases in these villages. Additionally, it could provide valuable insights for implementing Tafenoquine MDA on a larger scale.

ELIGIBILITY:
Inclusion Criteria:

* All village residence, aged >6 months who agrees to participate in the research.

Exclusion Criteria:

* People who refuse to participate
* People who are hypersensitive to Tafenoquine or Chloroquine
* Critically ill patient

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1242 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs) to assess safety and tolerability of Tafenoquine MDA | Baseline survey to end of Month-1 survey
  Number of (serious) adverse events reported

SECONDARY OUTCOMES:
To compare the incidence by Rapid Diagnostic Test (RDT) of P. vivax before and 1-3-6 months after providing the single round of MDA with Tafenoquine radical cure treatment | Month 1, 3 and 6
  Malaria Incidence by RDT reported from malaria post at month 1, 3 and 6
To evaluate the adherence of healthcare workers to the SOP for implementing MDA of Tafenoquine. | Baseline survey and Month-1 survey
  Proportion of village health workers adhere to the SOP for G6PD testing & documentation, tafenoquine administration and adverse event recording & reporting.
To compare the prevalence by PCR of P. vivax before and a month after providing the single round of MDA. | Baseline survey and Month-1 survey
  Difference in proportion positive to PCR positive before and a month after providing the single round of MDA.

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Result] Cohen JM, Smith DL, Cotter C, Ward A, Yamey G, Sabot OJ, Moonen B. Malaria resurgence: a systematic review and assessment of its causes. Malar J. 2012 Apr 24;11:122. doi: 10.1186/1475-2875-11-122. PMID 22531245
- [Result] Jaramillo-Ochoa R, Sippy R, Farrell DF, Cueva-Aponte C, Beltran-Ayala E, Gonzaga JL, Ordonez-Leon T, Quintana FA, Ryan SJ, Stewart-Ibarra AM. Effects of Political Instability in Venezuela on Malaria Resurgence at Ecuador-Peru Border, 2018. Emerg Infect Dis. 2019 Apr;25(4):834-836. doi: 10.3201/eid2504.181355. Epub 2019 Apr 17. PMID 30698522
- [Result] Nguyen TN, von Seidlein L, Nguyen TV, Truong PN, Hung SD, Pham HT, Nguyen TU, Le TD, Dao VH, Mukaka M, Day NP, White NJ, Dondorp AM, Thwaites GE, Hien TT. The persistence and oscillations of submicroscopic Plasmodium falciparum and Plasmodium vivax infections over time in Vietnam: an open cohort study. Lancet Infect Dis. 2018 May;18(5):565-572. doi: 10.1016/S1473-3099(18)30046-X. Epub 2018 Feb 2. PMID 29398388
- [Result] Okell LC, Bousema T, Griffin JT, Ouedraogo AL, Ghani AC, Drakeley CJ. Factors determining the occurrence of submicroscopic malaria infections and their relevance for control. Nat Commun. 2012;3:1237. doi: 10.1038/ncomms2241. PMID 23212366
- [Result] Poonkham, J. (2022). A Paradise Lost in the Indo-Pacific? Great Power Politics and International Relations of the Myanmar Tragedy. In: Yamahata, C., Anderson, B. (eds) Demystifying Myanmar's Transition and Political Crisis. Palgrave Macmillan, Singapore. https://doi.org/10.1007/978-981-16-6675-9_11